CLINICAL TRIAL: NCT00371891
Title: The Ontario Multidetector Computed Tomography (MDCT) Coronary Angiography Study (OMCAS)
Brief Title: Ontario Multidetector Computed Tomographic (MDCT) Coronary Angiography Study (OMCAS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Ron Goeree, Programs for Assessment of Technology in Health (PATH) Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HTA007-0603-01
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Coronary Arteriosclerosis; Cardiomyopathies; Heart Defects, Congenital; Heart Valve Diseases
MeSH Terms: conditions — Coronary Artery Disease; Cardiomyopathies; Heart Defects, Congenital; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Multidetector Computed Tomography Coronary Angiography — 1 Multidetector Computed Tomography Coronary Angiography

SUMMARY:
Multidetector Computed Tomographic Coronary Angiography (MDCTCA) has been recently demonstrated to be accurate and may be used as a potential alternative to conventional invasive coronary angiography, which requires cardiac catheterization, for the diagnosis of coronary artery disease. The purpose of this study is to see if MDCTCA can identify significant coronary artery disease as good as or better than conventional coronary angiography (CICA). The study is designed to enroll 900 subjects and is being conducted in 6 hospitals in Ontario. Subjects scheduled for conventional cardiac catheterization and coronary angiography will receive an additional test using MDCTCA. The information gathered during the MDCTCA will be compared to the results of the scheduled conventional invasive coronary angiogram.

ELIGIBILITY:
Inclusion Criteria:

Group 1

* Valvular heart disease (mitral stenosis, mitral regurgitation, aortic stenosis or aortic insufficiency) or
* Congenital heart disease (i.e. VSD, ASD, PDA) or
* Cardiomyopathy OR

Group 2

* Intermediate probability of coronary artery disease (probability of 10-90%) after clinical evaluation and traditional non-invasive testing

Exclusion Criteria:

* Age < 18 years
* Lack of consent
* Renal Insufficiency (GFR < 60 mL/min)
* Allergy to contrast agent
* Refractory angina requiring urgent/emergent coronary angiography (as per treating physician)
* Pregnancy or breast feeding
* Uncontrolled heart rate
* Previous CABG or PCI/Stent
* Chronic atrial fibrillation
* History of acute myocardial infarction, as defined by a creatine kinase (CK) level greater than 2 times normal with a troponin level above 4.
* Unable to perform 20 second breath-hold

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2006-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of MDCTCA as compared to CICA | After both MDCTCA and CICA are completed

SECONDARY OUTCOMES:
Descriptive statistics (rates and proportions) will be calculated for the number of "avoidable" diagnostic cardiac catheterizations. | After both MDCTCA and CICA are completed
The accuracy of MDCTCA to CICA will be compared in categorizing patients inot single, double, triple vessel, left main disease or no coronary stenosis. | After both MDCTCA and CICA are completed
The accuracy of MDCTCA to eliminate correctly the need for CICA will be calculated. | After both MDCTCA and CICA are completed

CONTACTS AND LOCATIONS:
Overall Officials: Michael Freeman, MD, Study Chair — Unity Health Toronto; Alan Moody, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Benjamin Chow, MD, Principal Investigator — Ottawa Heart Institute Research Corporation; Ronald Goeree, MA, Study Chair — Program for Assessment of Technology in Health, St. Joseph's Healthcare/McMaster University; Narinder Paul, MD, Principal Investigator — University Health Network, Toronto
Locations (4):
- Canada (4):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario

REFERENCES:
- [Derived] Chow BJ, Freeman MR, Bowen JM, Levin L, Hopkins RB, Provost Y, Tarride JE, Dennie C, Cohen EA, Marcuzzi D, Iwanochko R, Moody AR, Paul N, Parker JD, O'Reilly DJ, Xie F, Goeree R. Ontario multidetector computed tomographic coronary angiography study: field evaluation of diagnostic accuracy. Arch Intern Med. 2011 Jun 13;171(11):1021-9. doi: 10.1001/archinternmed.2011.74. Epub 2011 Mar 14. PMID 21403014